CLINICAL TRIAL: NCT01484951
Title: Assessing the Safety and Efficacy of Switching to AZARGA® (Brinzolamide/Timolol Fixed Combination) as Replacement Therapy in Patients With Uncontrolled Intraocular Pressure in Taiwan
Brief Title: AZARGA Transition Study in Taiwan for Patients With Uncontrolled Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-10-11
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Glaucoma
Keywords: Open-angle glaucoma; Ocular hypertension; Pigment dispersion glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Timolol; Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZARGA (Experimental): Brinzolamide 1% and timolol 0.5% fixed combination eye drops, one drop administered to the study eye(s) twice daily (8:00 am and 8:00 pm) for up to 8 weeks.
  Interventions: Drug: Brinzolamide 1% and timolol 0.5% fixed combination eye drops

INTERVENTIONS:
Drug: Brinzolamide 1% and timolol 0.5% fixed combination eye drops
  Other Names: AZARGA®

SUMMARY:
The purpose of this study was to assess the safety and efficacy of switching to Azarga from prior pharmacotherapy in patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in both eyes.
* Must be on a stable regimen of intra-ocular pressure (IOP) lowering medication within one week of screening/baseline visit.
* Must have an IOP of between 19 and 35 mmHg (both inclusive) in at least one eye, which would be the study eye, at screening.
* Must be willing to discontinue the use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study.
* Must have best corrected visual acuity of 6/60 (20/200 Snellen, 1.0 LogMAR) or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of the medication to be used in the study deemed clinically significant in the opinion of the principal investigator.
* Any abnormality preventing reliable applanation tonometry in either eye.
* Risk of visual field or visual acuity worsening as a consequence of participating in this study, in the investigator's best judgment.
* Pregnant or lactating.
* Participation in any other investigational study within 30 days of screening visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 study centers in Taiwan.
Period: Overall Study
Arm/Group | AZARGA
Started | 74
Completed | 69
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Personal Reasons | 1
Not completed — Non-Compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | AZARGA
Number analyzed (Participants) | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 32
Region of Enrollment [Number; unit: participants]
  Taiwan | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) at the Final Visit From Prior Beta-blocker Monotherapy (Timolol 0.5% Only)
Description: As measured at baseline and final visit with Goldmann applanation tonometry. The outcome measure was pre-specified for Timolol 0.5% only participants.
Time Frame: Baseline, Week 8
Population: Per protocol: All participants who received study medication, completed all study visits, and satisfied inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | AZARGA
Number analyzed (Participants) | 9
millimeters mercury (mmHg)
  Baseline | 18.22 (2.64)
  Change at Week 8 | -3.56 (3.16)

2. Secondary Outcome: Percentage of Patients With Target IOP (≤18 mmHg), Regardless of Prior Therapy
Description: As measured with Goldmann applanation tonometry. The outcome measure was pre-specified for all participants.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | AZARGA
Number analyzed (Participants) | 70
Percentage of Participants | 54.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (e.g., 10 months, 8 days). Individual adverse events were captured from the time of first administration of test article to the end-of-study visit (8 weeks).
Arm/Group | AZARGA
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 5/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZARGA (N=74)
Vision blurred (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right to review the results communication prior to its public release.